CLINICAL TRIAL: NCT01067729
Title: A Multi-Center, Randomized, Prospective Study of the Treatment of Superficial Partial-Thickness Burns: AWBAT™ vs. Biobrane®
Brief Title: A Postmarket Randomized Study of the Treatment of Superficial Partial-Thickness Burns Using Two Dressings
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Aubrey Inc. (Industry)
Responsible Party: Stephen Moss/President, Aubrey Inc.
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #AW-101508MC
Record Dates: First submitted 2010-02-10; First posted 2010-02-12 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2010-02

CONDITIONS: Burns
Keywords: Burn; Superficial burns; Partial thickness burns; Rate of healing; Infection rate; Pain perception; Non adherence; Scarring
MeSH Terms: conditions — Burns; Cicatrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: AWBAT Wound Dressing
  Other Names: Biobrane
Device: AWBAT™, Biobrane® — Comparison of burn dressings on randomized body sites using patient as own control

SUMMARY:
The purpose of this research study is to compare the rate of healing, the infection or complication rate, pain perception and scarring from burn injuries using two types of burn dressings.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate AWBAT™ compared to Biobrane® for the treatment of superficial partial-thickness burns using the patient as their own control.

ELIGIBILITY:
Inclusion Criteria:

* Superficial partial thickness burns
* Two non-contiguous burn sites or the same approximate size/depth for comparison, OR
* One burn site large enough to accommodate both a 6" square AWBAT™ dressing and a 6 " square Biobrane® dressing
* Burn wounds measuring >2% - <40% TBSA
* Patient age: >1 - 70 years

Exclusion Criteria:

* Ventilator dependence
* Pregnancy/Lactation
* Mechanism of injury was electrical, chemical or frostbite
* Co-morbidity which may compromise healing
* Known allergy to porcine or porcine products

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Dates: Start 2009-11; Primary Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Rate of healing | Day 14

SECONDARY OUTCOMES:
Scarring | 6 months, 1 year, 18 months and 2 years

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - UC Irvine Burn Center, Irvine, California
  - University of Missouri Health Care, Columbia, Missouri
  - Shriners Hospitals for Children, Galveston, Texas